CLINICAL TRIAL: NCT02443246
Title: A Prospective, Multi-centre, Randomized, Double-blind, Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of Vitamin D3 B.O.N. Intramuscular Injection in Adults With Vitamin D Deficiency
Brief Title: A Prospective, Multi-center Study to Evaluate the Efficacy and Safety of Vitamin D3 B.O.N. Intramuscular Injection in Adults With Vitamin D Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kwang Dong Pharmaceutical co., ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KDBON-302
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D deficiency (Experimental): Group 1
  Interventions: Drug: Vitamin D3 B.O.N. Injection (cholecalciferol 200,000IU); Drug: Placebo
- Vitamin D deficiency (Low) (Experimental): Group 2
  Interventions: Drug: Vitamin D3 B.O.N. Injection (cholecalciferol 200,000IU); Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 B.O.N. Injection (cholecalciferol 200,000IU)
Drug: Placebo

SUMMARY:
To compare the efficacy of Vitamin D3 B.O.N. Intramuscular Injection within 12 weeks with that of placebo in adults with Vitamin D Deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with vitamin D deficiency

Exclusion Criteria:

* Subjects who experienced a hypersensitivity to the cholecalciferol
* Subjects with renal impairment
* Subjects with Hypercalcemia
* Subjects with Hypercalciuria
* Subjects with clinically doubted calcium stone
* Subjects diagnosed with sarcoidosis
* Subjected diagnosed with pseudo-hypoparathyroidism
* Subjected with malignancy
* Subjects with clinically significant cardiovascular or lung impairment Judged by the investigator
* Subjects with the below laboratory abnormality (Platelet, WBC, Absolute neutrophil count, Albumin, AST or ALT)
* Subjects who are to take vitamin D supplements during the study period

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoints (serum 25(OH)D concentration) | 12 weeks
  serum 25(OH)D concentration

SECONDARY OUTCOMES:
Secondary Efficacy Endpoints (serum 25(OH)D concentration) | 24 weeks
  serum 25(OH)D concentration

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Kil Lim, Professor, Principal Investigator — Severance Hospital Seoul, Korea; Yun-seok Jeong, Professor, Principal Investigator — Ajou University Hospital, Korea; Han-seok Choi, Professor, Principal Investigator — Dongguk University Ilsan Hospital, Korea